CLINICAL TRIAL: NCT00779805
Title: An Open Label, Balanced, Randomised, Two-Treatment, Two-Period, Two-Sequence, Single-Dose, Crossover Bioavailability Study on Pseudoephedrine Hydrochloride Formulations Comparing Pseudoephedrine Hydrochloride 120 mg ER Tablets of Ranbaxy Laboratories With Sudafed 120 mg ER Tablets of Pfizer Consumer Health Care in Healthy, Adult, Human Subjects Under Fed Conditions.
Brief Title: Bioequivalence Study of Pseudoephedrine HCl 120 mg ER Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 016/ PSEUD-120/ 04
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence Pseudoephedrine hydrochloride 120 mg ER tablets
MeSH Terms: interventions — Pseudoephedrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Pseudoephedrine hydrochloride 120 mg ER tablets of Ranbaxy
  Interventions: Drug: Pseudoephedrine hydrochloride 120 mg ER tablets
- 2 (Active Comparator): Sudafed 120 mg ER tablets
  Interventions: Drug: Pseudoephedrine hydrochloride 120 mg ER tablets

INTERVENTIONS:
Drug: Pseudoephedrine hydrochloride 120 mg ER tablets

SUMMARY:
The objective of the study was to compare the single dose oral bioavailability of Pseudoephedrine hydrochloride 120 mg ER tablets of Ranbaxy with Sudafed 120 mg ER tablets of Pfizer Consumer Health Care in healthy, adult, human subjects under fed conditions.

DETAILED DESCRIPTION:
This study was an open label, balanced, randomized, two-treatment, two-period, two-sequence, single dose crossover bioavailability study planned on 40 healthy, adult, human subjects under fed conditions.

A total of forty (40) healthy, adult, human subjects were admitted in the study to allow the dosing in the first period. Out of the forty subjects, only thirty eight (38) subjects completed both the periods of the study.

ELIGIBILITY:
Inclusion Criteria:

* Be in the age range of 18 - 45 years
* Be neither over weight nor under weight for his/ her height as per the Life Insurance Corporation of India height/ weight chart for non-medical cases
* Have voluntarily given written informed consent to participate in this study
* Be of normal health as determined by medical history and physical examination of the subjects performed within 14 days prior to the commencement of the study
* If female and:
* Of child bearing potential is practicing an acceptable method of birth control for the duration of the study as judged by the investigator (s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence; or
* Is postmenopausal for at least 1 year; or
* Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)

Exclusion Criteria:

* History of allergy to Pseudoephedrine or other sympathomimetic drugs
* History of intake of any sympathomimetic drugs and glucocorticoids during a period of 15 days prior to day 1 of this study.
* Concurrent use of monoamine oxidase inhibitor (MAOI) drugs within 14 days prior to day 1 of this study
* Any evidence of organ dysfunction or any clinically significant deviations from the normal, in physical or clinical determinations
* Presence of disease markers of HIV 1 or 2, hepatitis B or C viruses or syphilis infection
* Female volunteers demonstrating a positive pregnancy test
* Female volunteers who are currently breastfeeding
* Presence of values which are significantly different from normal reference ranges (as defined in appendix 5) and/ or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol
* Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/ HPF), glucose (positive) or protein (positive)
* Clinically abnormal ECH or chest X-ray
* History of serious gastrointestinal, hepatic, renal, pulmonary, neurological or hematological diseases or glaucoma
* History of cardiovascular disorders (including hypertension), endocrine disorders, hyperthyroidism, diabetes mellitus, prostatic hypertrophy, palpitations, insomnia, tremors or bronchial asthma
* History of any psychiatric illness which may impair the ability to provide written informed consent
* Regular smokers who smoke more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
* History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or have difficulty in abstaining for the duration of each study period
* Use of any enzyme modifying drugs within 30 days prior to day 1 of this study
* Participation in any clinical trail within 12 weeks preceding day 1 of this study
* Subjects who, through completion of this study, would have donated and / or lost more than 350 mL of blood in the past 3 months.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2004-06; Primary Completion 2004-06 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Ranbaxy CPU, Gurgaon, Haryana, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html